CLINICAL TRIAL: NCT00730756
Title: A Pilot, Randomised, Double-blind, Placebo-controlled, Parallel-group, Multicentre Study to Evaluate the Efficacy and Safety of Once-daily Intranasal Administration of Fluticasone Furoate Nasal Spray 110 mcg for 4 Weeks in Adults and Adolescents With Irritant (Non-Allergic) Rhinitis
Brief Title: A Pilot Study In Adults And Adolescents With Irritant (Non-Allergic) Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR111158
Record Dates: First submitted 2008-02-27; First posted 2008-08-08 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Adolescents; Irritant(non-allergic)rhinitis; Adults; GW685698; Air Pollution
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A (Active Comparator): Fluticasone Furoate Nasal Spray 110mcg intranasally once daily
  Interventions: Drug: Fluticasone Furoate Nasal Spray
- Arm B (Placebo Comparator): Matching placebo nasal spray intranasally once daily
  Interventions: Other: Placebo Nasal Spray

INTERVENTIONS:
Drug: Fluticasone Furoate Nasal Spray — Fluticasone furoate nasal spray 110mcg intranasally once daily for 4 weeks
  Other Names: GW685698
  Arms: Arm A
Other: Placebo Nasal Spray — Matching placebo nasal spray intranasally once daily for 4 weeks
  Arms: Arm B

SUMMARY:
The purpose of this pilot study is to compare the effects (effectiveness and safety)of an intranasal corticosteroid (fluticasone furoate nasal spray [FFNS]) with a placebo nasal spray for the treatment of irritant (non-allergic) rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Subject is willing and able to provide consent to participate in the study. For subjects who are under 18 years of age, an appropriately signed and dated assent must be obtained from the parents or guardian.
* Outpatient: Subject is treatable on an outpatient basis.
* Age: 12 years of age or older at Visit 2.
* Gender: Male or eligible female

To be eligible for entry into the study, females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control, as defined by the following:

* Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
* Implants of levonorgestrel
* Injectable progestogen
* Oral contraceptive (either combined estrogen/progestin or progestin only)
* Any intrauterine device (IUD) with a documented failure rate of less than 1% per year, or
* Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days).
* Double barrier method - spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a spermicide and female diaphragm).

Female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A urine pregnancy test will be performed at the screening visit (Visit 1), the randomisation visit (Visit 2) and at the final visit (Visit 6 or Early Withdrawal).

* Clinical history: Diagnosis or evidence of air pollution triggers as the predominant irritant trigger for their rhinitis symptoms to include ALL of the following:

  * A two year clinical history of irritant (non-allergic) rhinitis triggered predominantly by air pollution exposure (written or verbal confirmation) in the opinion of the investigator and evidence of symptoms such as rhinorrhea, nasal congestion and postnasal drip relating to concentration of air particulates, air quality and levels of exposure.
  * Based on the trigger questionnaire, subjects must indicate that air pollution is the predominant trigger that makes their rhinitis symptoms worse completed at Visit 1.
  * Negative skin test (by prick method) response to seasonal allergens (including tree, grass and weed pollens) and perennial allergens (including animal dander, house dust mites, cockroach and mould) relevant to the geographical area completed at Visit 1.

A negative response for allergen skin prick testing is defined as a wheal <3 mm than the diluent control.

* Positive response to a histamine skin test (prick method) completed at Visit 1. A positive response for histamine skin prick testing is defined as a wheal ≥3 mm larger than the diluent control.
* Normal sinus radiograph (Waters view) to rule out sinusitis (presence of mucosal thickening of ≥6 mm at the point of maximal thickening or an air fluid level or opacification). The sinus radiograph will be scheduled at Visit 1.

  * Ability to comply with study procedures: Subject understands and is willing, able and likely to comply with study procedures and restrictions.
  * Literate: Subject must be able to read, comprehend, and record information in English or native language.

Randomization Criteria

* Average of the last 8, reflective, total nasal symptom score (rTNSS) assessments (4 morning [AM] assessments, 4 evening [PM] assessments) over the four 24-hour periods prior to randomisation must be greater than/equal to 4.5.
* Average of the last 8 reflective nasal symptom assessments for congestion (4 AM assessments, 4 PM assessments) over the four 24-hour periods prior to randomisation must be greater than/equal to 2.
* A subject must have completed 80% of assessments on the screening symptom diary card.

Exclusion Criteria:

* Significant concomitant medical conditions, defined as but not limited to:

  * a historical or current evidence of clinically significant uncontrolled disease of any body system (e.g., tuberculosis, psychological disorders, eczema). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or which would confound the interpretation of the study results if the disease/condition exacerbated during the study.
  * a severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or nasal septal perforation that could affect the deposition of double blind intranasal study drug
  * nasal (e.g., nasal septum) or ocular injury/surgery in the last 3 months
  * asthma, with the exception of mild intermittent asthma [Global Initiative for Asthma (GINA), 2006]. NOTE: Subjects will be allowed to use short-acting inhaled beta2 agonists ONLY on an as needed basis.
  * rhinitis medicamentosa
  * bacterial or viral infection (e.g., common cold) of the upper respiratory tract within two weeks of Visit 1 or during the screening period
  * documented evidence of acute or significant chronic sinusitis, as determined by a sinus radiograph (Waters view) done at Visit 1
  * current or history of glaucoma and/or current cataract or ocular herpes simplex
  * physical impairment that would affect the subject's ability to participate in the study
  * clinical evidence of a Candida infection of the nose or oropharynx
  * history of psychiatric disease, intellectual deficiency, poor motivation, substance abuse (including drug and alcohol) or other conditions that will limit the validity of informed consent or that would confound the interpretation of the study results
  * history of or current use of cocaine
  * history of adrenal insufficiency
  * Chickenpox or measles within 3 weeks of Visit 1. A subject is not eligible if he/she currently has chickenpox or measles, or has been exposed to chickenpox or measles during the last 3 weeks and is non-immune. If a subject develops chickenpox or measles during the study, he/she will be withdrawn from the study. If a non-immune subject is exposed to chickenpox or measles during the study, his/her continuation in the study will be at the discretion of the investigator, taking into consideration the likelihood of developing active disease.
* Use of corticosteroids, defined as:

  * Intranasal corticosteroid within 4 weeks prior to Visit 1.
  * Inhaled, oral, intramuscular, intravenous, ocular, and/or dermatological corticosteroid (with the exception of hydrocortisone cream/ointment, 1% or less, or equivalent) within 8 weeks prior to Visit 1.
* Use of other allergy medications within the timeframe indicated relative to Visit 1

  * Intranasal or ocular cromolyn within 14 days prior to Visit 1
  * Short-acting prescription and over the counter (OTC) antihistamines, including ocular preparations and antihistamines contained in insomnia and 'nighttime' pain formulations taken for insomnia, within 7 days prior to Visit 1
  * Long-acting antihistamines within 10 days prior to Visit 1: loratadine, desloratadine, fexofenadine, cetirizine
  * Long-acting antihistamine, astemizole, within 12 weeks prior to Visit 1
  * Intranasal antihistamines (e.g. Astelin) within 2 weeks prior to Visit 1
  * Oral or intranasal decongestants within 3 days prior to Visit 1
  * Intranasal, oral, or inhaled anticholinergics within 3 days prior to Visit 1
  * Oral antileukotrienes within 3 days prior to Visit 1
  * Subcutaneous omalizumab (Xolair) within 5 months of Visit 1
  * Use of any medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole.
  * Ocular antihistamines, artificial tears, eyewashes/nasal irrigation solutions, homeopathic preparations, lubricants, sympathomimetic or vasoconstrictor preparations during the screening or treatment periods. No exclusion period prior to screening (Visit 1) is required for these treatments.
  * Throat treatments (e.g., cough lozenges, throat sprays) during the screening and treatment periods. No exclusion period prior to screening (Visit 1) is required for these treatments.
* Use of other medications that may affect irritant rhinitis or its symptoms

  * Chronic use of concomitant medications, such as tricyclic antidepressants, that would affect assessment of the effectiveness of the study drug.
  * Chronic use of long-acting beta-agonists (e.g., salmeterol).
  * Chronic use of other intranasally administered medications (e.g., calcitonin-salmon).
  * Use of face masks (e.g, general face masks that are used for protection from air pollution, and C-PAP face masks or pillows), saline nasal sprays and lavages, eye drops, and local, herbal and homeopathic treatments.
* Chronic use of medications that could cause drug-induced rhinitis including:

  * ACE inhibitors, reserpine, guanethidine, methyldopa, hydralazine, beta-blockers, alpha-adrenoceptor antagonists (e.g., Prazosin), phentolamine, chlorpromazine, aspirin, and non-steroidal anti-inflammatory medications (NSAIDS).

NOTE: Subjects taking aspirin and/or NSAIDs on a chronic basis may be considered for inclusion in the study if the investigator can evaluate and document the subject's irritant rhinitis symptoms are not caused by these medications.

* Use of immunosuppressive medications 8 weeks prior to screening and during the study
* Immunotherapy
* Allergy/Intolerance

  • Known hypersensitivity to corticosteroids, or any excipients in the product
* Clinical trial/experimental medication experience

  * Exposure to an investigational study drug within 30 days prior to Visit 1
  * Participation in a previous or current fluticasone furoate nasal spray (GW685698X) clinical study
* Positive or inconclusive pregnancy test or female who is breastfeeding

  • Has a positive or inconclusive pregnancy test at Visit 1 or Visit 2
* Tobacco use

  • Subjects who currently use or have used within the past year smoking products including cigarettes, cigars and pipes, or smokeless products such as chewing tobacco.
* Findings of a clinically significant, abnormal electrocardiogram (ECG)
* Findings of a clinically significant laboratory abnormality

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tantilipikorn P, Thanaviratananich S, Chusakul S, Benjaponpitak S, Fooanant S, Chintrakarn C, Jirapongsananuruk O, Visitsunthorn N, Toler T, Sutton L, Wu W, Lee L. Efficacy and Safety of Once Daily Fluticasone Furoate Nasal Spray for Treatment of Irritant (Non-allergic) Rhinitis. Open Respir Med J. 2010 Nov 3;4:92-9. doi: 10.2174/1874306401004010092. PMID 21253453
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR111158 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Vehicle placebo nasal spray once daily
- FFNS 110 mcg: Fluticasone Furoate Nasal Spray (FFNS) 110 micrograms (mcg) once daily
Period: Overall Study
Arm/Group | Placebo | FFNS 110 mcg
Started | 49 | 53
Completed | 45 | 48
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Deviation | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrew Consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FFNS 110 mcg | Total
Number analyzed (Participants) | 49 | 53 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants must have been 12 years of age or older.
  years | 35.9 (10.89) | 37.1 (12.78) | 36.6 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 12 | 20 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 49 | 53 | 102
Total Nasal (TNSS) and Total Ocular (TOSS) Symptom Scores [Mean (Standard Deviation); unit: points on a scale] — Total Symptom Scores (scale of 0-9; sum of the three individual nasal or ocular scores) based on 3 nasal symptoms (rhinorrhea, nasal congestion, and post-nasal drip) and 3 ocular symptoms (eye itching/burning, eye tearing/watering, and eye redness). Symptoms were evaluated on a scale of 0 (none), 1 (mild), 2 (moderate), or 3 (severe).
  points on a scale
    Daily Reflective TNSS | 6.4 (1.16) | 6.7 (1.25) | 6.5 (1.22)
    Morning (AM) pre-dose instantaneous (i) TNSS | 6.3 (1.50) | 6.5 (1.57) | 6.4 (1.53)
    AM Reflective TNSS | 6.4 (1.24) | 6.7 (1.36) | 6.5 (1.30)
    Evening (PM) Reflective TNSS | 6.3 (1.31) | 6.7 (1.32) | 6.5 (1.32)
    Daily Reflective TOSS | 2.4 (2.17) | 3.1 (2.27) | 2.8 (2.24)
    AM pre-dose iTOSS | 2.4 (2.24) | 3.1 (2.17) | 2.8 (2.22)
    AM Reflective TOSS | 2.4 (2.20) | 3.0 (2.16) | 2.7 (2.19)
    PM Reflective TOSS | 2.4 (2.19) | 3.2 (2.42) | 2.8 (2.34)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daily rTNSS Over the Entire Treatment Period (28 Days)
Description: The Total Nasal Symptom Score (TNSS) is the sum (scale 0-9) of the individual nasal scores for rhinorrhea, nasal congestion, and post-nasal drip. All symptoms were evaluated using a scale of 0 (None), 1 (Mild), 2 (Moderate), or 3 (Severe). Reflective (r) assessments were performed in the morning (AM) and evening (PM) and assessed the participant's symptoms over the preceding 12 hours. The daily reflective Total Nasal Symptoms Score (daily rTNSS) is the average of the AM and PM rTNSS. Mean change from baseline was calculated as the participant's treatment period mean minus the baseline mean.
Time Frame: Baseline through Week 4 (28 days)
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale | -2.10 (0.25) | -2.17 (0.23)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg; Test type: Superiority or Other; p = 0.845, ANCOVA; Center, baseline eosinophils, baseline symptom score, age, and gender were included as covariates in all efficacy analyses

2. Secondary Outcome: Mean Change From Baseline in AM rTNSS, PM rTNSS, and AM Pre-dose iTNSS Over the Entire Treatment Period (28 Days)
Description: The TNSS is the Total Nasal Symptom Score (scale 0-9), a sum of the individual nasal scores for (1) rhinorrhea, (2) nasal congestion, and (3) post-nasal drip. All 3 symptoms were evaluated using a scale of: 0 (None), 1 (Mild), 2 (Moderate), or 3 (Severe). Reflective (r) assessments were performed in the morning (AM) and evening (PM) and assessed the participant's symptoms over the preceding 12 hours (AM rTNSS, PM rTNSS). The AM pre-dose instantaneous assessment (AM pre-dose iTNSS) was performed in the morning just prior to dosing and assessed symptoms at that moment.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  AM pre-dose iTNSS | -1.82 (0.26) | -1.90 (0.24)
  AM rTNSS | -2.13 (0.27) | -2.15 (0.24)
  PM rTNSS | -2.09 (0.25) | -2.19 (0.23)

3. Secondary Outcome: Mean Change From Baseline in Daily Reflective Individual Nasal Symptoms Score Over the Entire Treatment Period (28 Days)
Description: Mean change for the individual symptoms of rhinorrhea, nasal congestion, and post-nasal drip. Reflective rating represents the participant's symptoms over the preceding 12 hours. Reflective assessments were performed in the morning (AM) and evening (PM). The daily reflective individual nasal symptom score average of the AM and PM reflective individual nasal symptoms is the daily reflective individual nasal symptom score. All symptoms were evaluated on a 0 (none) to 3 (severe) scale.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  Rhinorrhea | -0.64 (0.09) | -0.72 (0.08)
  Nasal congestion | -0.75 (0.09) | -0.79 (0.08)
  Post-nasal drip | -0.70 (0.10) | -0.67 (0.09)

4. Secondary Outcome: Mean Change From Baseline in AM Pre-dose Instantaneous Individual Nasal Symptoms Over the Entire Treatment Period (28 Days)
Description: The AM pre-dose instantaneous assessment is performed in the morning prior to dosing and evaluates symptoms at that moment. The individual symptoms of rhinorrhea, nasal congestion, and post-nasal drip were measured at this time. All three symptoms were evaluated using a 0 (none) to 3 (severe) scale. This assessment provides information on the duration of action of the treatment.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  Rhinorrhea | -0.52 (0.09) | -0.61 (0.09)
  Nasal congestion | -0.64 (0.09) | -0.71 (0.08)
  Post-nasal drip | -0.66 (0.10) | -0.58 (0.09)

5. Secondary Outcome: Mean Change From Baseline in AM and PM Reflective Individual Nasal Symptoms Over the Entire Treatment Period (28 Days)
Description: Mean change for the individual symptoms of rhinorrhea, nasal congestion, and post-nasal drip as measured in the morning and evening. Reflective rating represents the participant's symptoms over the preceding 12 hours. All symptoms were evaluated on a 0 (none) to 3 (severe) scale.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  AM, rhinorrhea | -0.65 (0.09) | -0.72 (0.08)
  PM, rhinorrhea | -0.63 (0.09) | -0.72 (0.09)
  AM, nasal congestion | -0.75 (0.09) | -0.78 (0.08)
  PM, nasal congestion | -0.76 (0.09) | -0.79 (0.09)
  AM, post-nasal drip | -0.73 (0.10) | -0.65 (0.09)
  PM, post-nasal drip | -0.69 (0.10) | -0.68 (0.09)

6. Secondary Outcome: Mean Change From Baseline in Total Ocular Symptoms Over the Entire Treatment Period (28 Days)
Description: The Total Ocular Symptom Score (TOSS) is a sum (scale 0-9) of the individual ocular scores for eye itching/burning, eye tearing/watering, and eye redness. All 3 symptoms were evaluated using a scale of 0 (None), 1 (Mild), 2 (Moderate), or 2 (Severe). The daily reflective TOSS (daily rTOSS) is the average of the morning (AM) and evening (PM) rTOSS assessments that measure symptoms over the previous 12 hours. The AM pre-dose instantaneous (iTOSS) assessment is performed in the morning prior to dosing and evaluates symptoms at that moment, providing data on the duration of action of treatment.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  Daily rTOSS | -0.77 (0.16) | -1.04 (0.14)
  AM pre-dose iTOSS | -0.85 (0.17) | -0.98 (0.15)
  AM rTOSS | -0.81 (0.17) | -0.96 (0.16)
  PM rTOSS | -0.74 (0.16) | -1.13 (0.15)

7. Secondary Outcome: Mean Change From Baseline in Daily Reflective Individual Ocular Symptoms Over the Entire Treatment Period (28 Days)
Description: Mean change for the individual symptoms of eye itching/burning, eye tearing/watering, and eye redness. Reflective rating represents the participant's symptoms over the preceding 12 hours. Reflective assessments were performed twice daily (AM and PM). The average of the AM and PM reflective individual ocular symptoms is the daily reflective individual ocular symptoms. Reflective individual ocular symptoms were evaluated on a 0 (none) to 3 (severe) scale.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  Eye itching/burning | -0.32 (0.07) | -0.45 (0.06)
  Eye tearing/watering | -0.29 (0.06) | -0.31 (0.06)
  Eye redness | -0.17 (0.06) | -0.28 (0.05)

8. Secondary Outcome: Mean Change From Baseline in AM Pre-dose Instantaneous Individual Ocular Symptoms Over the Entire Treatment Period (28 Days)
Description: The AM pre-dose instantaneous assessment is performed in the morning prior to dosing and evaluates symptoms at that moment. The individual symptoms of eye itching/burning, eye tearing/watering, and eye redness were measured at this time. All three symptoms were evaluated using a 0 (none) to 3 (severe) scale. This assessment provides information on the duration of action of the treatment.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  Eye itching/burning | -0.35 (0.08) | -0.37 (0.07)
  Eye tearing/watering | -0.30 (0.06) | -0.33 (0.06)
  Eye redness | -0.21 (0.05) | -0.27 (0.05)

9. Secondary Outcome: Mean Change From Baseline in AM and PM Reflective Individual Ocular Symptoms Over the Entire Treatment Period (28 Days)
Description: Mean change for the individual symptoms of eye itching/burning, eye tearing/watering, and eye redeness. Reflective ratings assessed the participant's symptoms over the preceding 12 hours. Reflective assessments were performed twice daily (AM and PM) and were evaluated on a 0 (none) to 3 (severe) scale.
Time Frame: Baseline through Week 4 (28 days)
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | FFNS 110 mcg
Number analyzed (Participants) | 49 | 53
points on a scale
  AM, eye itching/burning | -0.34 (0.07) | -0.42 (0.06)
  PM, eye itching/burning | -0.30 (0.07) | -0.48 (0.06)
  AM, eye tearing/watering | -0.32 (0.07) | -0.29 (0.06)
  PM, eye tearing/watering | -0.27 (0.06) | -0.33 (0.05)
  AM, eye redness | -0.16 (0.06) | -0.23 (0.05)
  PM, eye redness | -0.19 (0.06) | -0.31 (0.05)

ADVERSE EVENTS:
Arm/Group | Placebo | FFNS 110 mcg
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/53
Other Adverse Events (participants affected / at risk) | 3/49 | 9/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | FFNS 110 mcg (N=53)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | FFNS 110 mcg (N=53)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Migraine (Nervous system disorders) | 1 | 2
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.